CLINICAL TRIAL: NCT06959238
Title: Investigation of the Effects of Basic Body Awareness Therapy on Core Muscle Endurance, Posture, Balance, Quality of Life and Body Awareness in Earthquake Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: Cumhuriyet University (Other); Gazi University (Other)
Responsible Party: Principal Investigator, Emine Nacar, Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/04-31
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Earthquake; Core; Posture; Balance; Quality of Life; Body Awareness
Keywords: Earthquake; core; posture; balance; quality of life; body awareness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Basic body awareness therapy (Active Comparator): Individuals in the intervention group will receive basic body awareness therapy (TBFT).The flow of an exercise session of TBFT is 10 minutes of body scan, 35 minutes of exercises and 15 minutes of feedback. TBFT exercises are performed on the back, sitting and standing with diaphragmatic breathing and the sound "m". The sound "m" is a universal sound and is used during all exercises. In addition, using the sound "m" during the exercises contributes positively to the respiratory functions of the participant as it creates resistance on the diaphragm. Participants catch the rhythm of breathing and movement by making the sound "m". A mat cushion is used for the exercises performed in the supine position, and a fixed stool with a hard surface suitable for the participants' leg length is used for the exercises performed in the sitting position. Exercises performed in the standing position are performed without shoes and on a hard surface.
  Interventions: Other: Temel beden farkındalığı terapisi
- Control group (No Intervention): Participants in the control group will not receive any intervention.

INTERVENTIONS:
Other: Temel beden farkındalığı terapisi — Individuals in the TBFT group will receive a total of 16 exercise sessions, with individual exercises 2 days a week for the first 2 weeks and group exercises 2 days a week for the next 6 weeks. The purpose of the individual sessions is to aim for the participant to learn the TBFT exercises and to prepare the participant for the group sessions. In individual sessions, the person learns body scanning and develops awareness about their own body. The participant continues the exercises they learned in the individual session at home. At this stage, the participant is assigned a notebook and is asked to write down their experiences of the exercises they do at home in this notebook. The participant who completes the individual sessions continues with the group sessions. The purpose of the group sessions is to provide interaction within the group and to establish a bond of trust between the individuals in the group with the interaction obtained. The fact that the participants do exercises toge
  Arms: Intervention group: Basic body awareness therapy

SUMMARY:
Earthquakes are natural disasters that occur unexpectedly, affecting many people negatively, threatening life and causing serious losses. In our geography where earthquakes are frequently experienced, two earthquakes occurred on February 6, 2023 in the Southeastern part of our country, the first with a magnitude of 7.7 and the second with a magnitude of 7.5. The earthquakes that occurred with Pazarcık/Kahramanmaraş as the epicenter are one of the major earthquakes in our country. It is known that a significant portion of individuals exposed to such large earthquakes are affected mentally and physically. However, although psychological effects have been known for many years, the physical changes that occur due to psychological effects are still being investigated today. Many studies on the subject focus on complaints of dizziness and disturbances in balance following an earthquake. However, it is also possible that different physical effects may develop. The aim of our current project proposal is to examine the effects of basic body awareness therapy on core muscle endurance, posture, balance, quality of life and body awareness in earthquake survivors. Within the scope of our project, 30 earthquake survivors between the ages of 18-45 who experienced the February 6, 2023 earthquake will be included in the study. For all individuals, evaluation of core muscles will be performed with McGill Endurance test, Prone Bridge test and Stabilizer Pressure Biofeedback, posture evaluation with New York Posture Assessment Method (NYPAM) and lateral digital imaging in standing posture, balance evaluation with Balance on One Leg test (eyes open and closed), Functional Forward Reach Test and Y Balance Test, quality of life evaluation with Short Form-36 (SF-36) and body awareness evaluation with Body Awareness Questionnaire (BAQ). Individuals will be divided into 2 groups by closed envelope randomization method. The first group was determined as the intervention group and the second group as the control group. While Basic Body Awareness Therapy will be applied to the individuals in the intervention group, no application will be made to the individuals in the control group. All assessments will be applied to individuals in both the intervention group and the control group 2 times in total at the beginning of the study and at the end of 8 weeks. Our project, which is foreseen to be completed in 12 months, is planned to be carried out in 16 sessions, 2 days a week, 1 hour a day, for 8 weeks, and to give home exercise 2 days a week, 1 hour a day. The fact that the evaluations to be applied within the scope of the project proposal and the exercise approach to be used have not been applied on earthquake victims before gives our study originality. It has the potential to form the basis for future studies in the field of health related to earthquake victims.

ELIGIBILITY:
Inclusion Criteria:

* Having experienced the earthquake in the provinces affected by the earthquake with the epicenter of February 6, 2023, Pazarcık/Kahramanmaraş, and declared a state of emergency with a level 4 alarm (Kahramanmaraş, Malatya, Hatay, Adıyaman, Şanlıurfa, Gaziantep, Osmaniye, Kilis, Diyarbakır, Adana)
* Being between the ages of 18-45
* Volunteer to work
* Being able to speak Turkish

Exclusion Criteria:

* Refusing to participate in the study at any stage
* Presence of communication problems (vision, hearing and speech disorders)
* Presence of limitation and contracture in the lower extremity
* Having had an amputation
* Polypharmacy and antidepressant use
* Presence of a diagnosed disease related to the psychiatric, neurological and musculoskeletal system.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Trunk flexor test | From registration to the start of treatment.
  The trunk flexor test is performed with the trunk at 60° flexion and the knees and hips at 90° flexion. The arms are crossed over the chest and the individuals are asked to maintain this position for as long as possible.
Trunk extensor test | From registration to the start of treatment.
  The trunk extensor test is performed in a prone position on the treatment table. The pelvis, hips and knees are fixed to the treatment table up to the level of the anterior superior iliac spine. Individuals are asked to maintain a horizontal body position for as long as possible with their arms crossed on their chest.
The side bridge test | From registration to the start of treatment.
  The side bridge test is performed on the mat while lying on the side. While lifting the hips up on the mat, the body weight is supported only by the elbows and feet below. The tests are terminated when the positions are disrupted. The measurement results are recorded in seconds.
Prone Bridge Test | From registration to the start of treatment.
  Subjects are asked to lift their bodies up by placing their weight on their forearms and toes while lying face down with their elbows in a flexed position. The test is terminated when the position is disrupted. The measurement results are recorded in seconds.
Stabilizer Pressure Biofeedback Unit Usage | From registration to the start of treatment.
  Stabilizer Pressure Biofeedback Unit measures the contraction force of the deep trunk muscles transversus abdominis. Chattanooga Stabilizer will be used in the measurement to be taken in this study. The inflatable device is placed centrally under the abdomen with its lower edge at the level of the anterior superior iliac spine. Before the test, individuals are taught how to selectively contract the transversus abdominis muscle with the corset method. After the pressure of the manometer is set to 70 mmHg, individuals are asked to reduce the pressure by slowly contracting the transversus abdominis muscle with the abdominal corset technique without holding their breath and to maintain this contraction for 5 seconds. The test is terminated if the pressure increases exceed 70 mmHg during the measurement. The average pressure change at the end of three contractions is calculated.
Posture assessment | From registration to the start of treatment.
  The postures of the individuals participating in the study will be assessed using the "New York Posture Assessment Method (NYPDY)". The individual is asked to stand in a resting position and points are given by observational assessment according to the posture patterns shown in the table. In this assessment system, changes in posture that may occur in 13 different parts of the body are scored by monitoring them. Accordingly, if the individual's posture is correct, five (5) points are given, if it is moderately impaired, three (3) points are given, and if it is severely impaired, one (1) points are given. The maximum total score obtained as a result of the test is 65 and the minimum is 13. The standard assessment criteria developed for this test are determined as "very good" if the total score is ≥ 45, "good" if it is 40-44, "moderate" if it is 30-39, "poor" if it is 20-29, and "poor" if it is ≤ 19. It is stated in the literature that the use of real-time (simultaneous) scoring limits
Single-Legged Balance Test | From registration to the start of treatment.
  This is a test in which the time the individual stands on the right and left lower extremities in balance is measured in seconds and evaluates static balance. The balance test on one leg is performed by recording the time from the moment the individual starts standing on one leg until the first moment when postural stability is disrupted. Measurements are performed in two stages: eyes open and closed. For the test performed with eyes open, the individual is asked to lift one leg without touching the supporting leg, look straight ahead and maintain their balance. For the test performed with eyes closed, the individual is asked to close their eyes, lift one leg without touching the supporting leg and maintain their balance. 360 seconds is accepted as the upper limit for the completion of the test.
Functional Forward Reach Test | From registration to the start of treatment.
  The maximum distance that an individual can reach forward and sideways while standing upright is measured in centimeters. In order to measure the distance reached, a tape measure is placed on the wall at the height of the individual's shoulder. The individual stands with their arm flexed at 90 degrees and their fist closed, without touching the wall but close to it. The assessor marks the head of the individual's 3rd metacarpal on the wall and asks the individual to reach forward as far as they can without taking a step. The assessor marks the head of the individual's 3rd metacarpal on the wall again and measures the difference between the beginning and the end with the tape measure. 15 cm and below indicates a significantly increased risk of falling, and 15 to 25 cm indicates a moderate risk of falling. The validity and reliability of the test were performed by Weiner et al.
Y Balance Test | From registration to the start of treatment.
  A simple but reliable test used to measure dynamic balance. It is a dynamic test performed in a single-legged stance that requires strength, flexibility, core control and proprioception. It is used to evaluate physical performance and to demonstrate functional symmetry. The validity and reliability of the test were performed by Plisky et al. Y balance kit is used to perform the test. All measurements are performed for both extremities while the individual is barefoot, barefoot and with their hands on their waists. While one extremity of the individual remains fixed on the ground, the other extremity is asked to go to the maximum distance it can extend in the anterior, posteromedial and posterolateral directions and return to the starting point in a balanced manner. After six trials in each direction for both legs, the tests will be performed in 3 repetitions. The average of the tests will be taken for each direction and the ratio to the leg length will be recorded in centimeters.
Assessment of Quality of Life | From registration to the start of treatment.
  One of the most frequently used questionnaires in the literature for assessing quality of life is the SF-36. It has a generic criterion feature among quality of life scales and provides wide-ranging measurement. It was developed and put into use by the Rand Corporation in 1992. It consists of a total of 36 items and provides measurement of a total of 8 dimensions: physical function, physical role difficulty, pain, general health, vitality, social function, emotional role difficulty and mental health. Scoring is done between 0-100. The value of "100" indicates good health status, and the value of "0" indicates poor health status. Its validity and reliability in Turkish was done in 1999.
Body Awareness Assessment | From registration to the start of treatment.
  Body Awareness Questionnaire will be used. The original name of the questionnaire is Body Awareness Questionnaire (BAQ). It was developed by Stephanie A. Shields and her colleagues in 1989. It is a scale that includes items related to the individual's physiological, psychological, emotional and social awareness levels, as well as sleep disorders, differences between being sick and not being sick, and physical and mental reactions and estimation levels specific to specific situations related to body awareness. Turkish validity and reliability were conducted in 2017. It consists of 18 items and 4 subgroups. A high score obtained from the questionnaire means a high level of body awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data include participants' measurements and their specific thoughts about therapy.